CLINICAL TRIAL: NCT07377591
Title: A Phase 1 Clinical Study to Evaluate the Safety, Tolerability, Efficacy and Pharmacokinetics of HDM2006 Monotherapy in Patients With Advanced Solid Tumors
Brief Title: A Study of HDM2006 in Patients With Advanced Solid Tumor
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HDM2006-101; CTR20244285 (Registry Identifier: China Drug Trials Center (CDE))
Record Dates: First submitted 2026-01-11; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HDM2006 (Experimental): In dose escalation phase, participants will be administered escalating doses of HDM2006 at 50 mg QD, ~1000 mg QD, Oral administration within half an hour after a meal. In dose expansion phase, participants will be administered to recommended dose for expansion (RDE) of HDM2006, Oral administration within half an hour after a meal.
  Interventions: Drug: HDM2006

INTERVENTIONS:
Drug: HDM2006 — Oral administration within half an hour after a meal, QD

SUMMARY:
This is a first-in-human (FIH) study to evaluate the safety and preliminary efficacy of experimental drug HDM2006 in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1. The subjects understand and voluntarily (or legally authorized guardian) sign a written informed consent form (ICF) approved by the Institutional Review Board (IRB) or Independent Ethics Committee (IEC).

  2. Males or females aged ≥ 18 years old. 3. In the dose escalation phase, subjects must have histologically or cytologically confirmed advanced or metastatic solid tumors, who have experienced adequate standard treatment failure, intolerance to standard treatment, or lack of effective standard treatment.

  4. In the dose expansion phase, subjects must have histologically or cytologically confirmed advanced or metastatic specific types of tumors, who have experienced adequate standard treatment failure, intolerance to standard treatment, or lack of effective standard treatment. These include, but are not limited to, head and neck squamous cell carcinoma, renal cell carcinoma, cervix carcinoma, and other advanced solid tumors, as well as tumor types that showed efficacy signals (CR/PR) in the dose escalation phase.

  5. In the dose expansion phase, subjects are able to provide fresh or archival (within one year) tumor tissues at the time of screening and are willing to provide tumor tissue biopsy after administration of HDM2006 for baseline and post-treatment biomarker analysis.

  6. Eastern Cooperative Oncology Group Performance Status (ECOG-PS) score of 0 or 1 .

  7. Expected survival time > 3 months. 8. According to the Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1), subjects in phase 1a must have at least one evaluable lesion, and subjects in phase 1b must have at least one measurable lesion (a lesion located in areas previously treated with radiotherapy will not be considered a measurable lesion unless there is sufficient evidence to show clear imaging progression of the lesion after radiotherapy; biopsy lesions should be excluded for measurable lesions in subjects in phase 1b).

  9. The subject has good organ function as indicated by laboratory results at screening (no cytokine or other corrective medications are allowed within 14 days prior to laboratory tests at screening):Hematology: a) absolute neutrophil count ≥ 1.5 × 10^9/L (1500/mm3); b) platelet count ≥ 100 × 10^9/L (no platelet transfusion within 14 days prior to the investigation); c) hemoglobin ≥ 9.0 g/dL (no red blood cell transfusion within 30 days prior to the investigation); Liver: a) serum total bilirubin ≤ 1.5 × ULN; b) AST and ALT ≤ 3 × ULN (≤ 5 × ULN for subjects with tumor liver metastasis); c) serum albumin ≥ 30 g/L (no albumin transfusion within 21 days prior to investigation); Kidney: blood creatinine ≤ 1.5 × ULN; or creatinine clearance (CrCl) ≥ 50 mL/min (calculated by Cockcroft-Gault formula, see Appendix 4); Coagulation function: international normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN (unless the subject is receiving anticoagulant therapy, and the coagulation parameters [PT/INR and APTT] are within the expected range for anticoagulant therapy at screening).

  10. Women of childbearing potential (WOCBP) must be willing to use 2 adequate methods of contraception or barrier contraception plus hormonal contraception from the time of signing ICF until 6 months after the last dose of study treatment to prevent pregnancy or abstain from heterosexual activity throughout the study; male subjects must agree to take adequate contraceptive measures from the first dose of study treatment until 6 months after the last dose of study treatment .

  11. Subject are willing and able to complete scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

* 1. Subjects who are concurrently participating in another clinical study, unless it is an observational (non-interventional) clinical study or they are in the survival follow-up period of an interventional study.

  2. Subjects with the following treatments:
  1. Subjects who have received major surgery within 4 weeks prior to the first dose, excluding minor surgery, such as appendicitis surgery, tissue acquisition for tumor biopsy, etc.;
  2. Subjects who have received bone marrow (equivalent to pelvic bone marrow area) or extensive radiotherapy within 28 days prior to the first dose; subjects who have received local radiotherapy (e.g., thoracic and rib radiotherapy) within 7 days prior to the first dose of the study drug;
  3. Subjects who have previously received HPK1 inhibitor treatment. 3. Subjects who have history of active malignancies within the past 2 years, with the exception of tumors in this study and cured local tumors, such as basal cell carcinoma of skin, squamous cell carcinoma of skin, superficial bladder cancer, cervix carcinoma in situ, breast cancer in situ, etc.

     4. Subjects who have not recovered (i.e., recover to ≤ Grade 1 or baseline) from related AEs (such as alopecia, ≤ Grade 2 sensory neuropathy, or other ≤ Grade 2 AEs that do not pose a safety risk as judged by the investigator) resulting from previous treatments or other anti-tumor therapies.

     5. Subjects with unstable brain metastasis: subjects with central nervous system complications requiring emergency neurosurgery (e.g., surgery) (excluding those who have completed surgery for more than 7 days and whose complications have resulted in ≤ Grade 1 side effects); 6. Subjects with epilepsy requiring treatment; subjects with a history of psychotropic drug abuse and unable to abstain or have mental disorders (those who have abstained must meet an observation period without withdrawal reactions for at least 2 weeks).

     7. Subjects with any of the following cardiovascular diseases/symptoms/signs:

  a) Mean QTc (corrected QT interval, calculated by Fridericia's formula) at rest: male > 450 ms, female > 470 ms, with the mean QTc of triplicate ECG measurements within ≥ 5 min (at least 1 min interval between two measurements, QT interval measurement should be from the beginning of the QRS complex to the end of the T wave); b) Any important abnormalities with clinically significant in rhythm, conduction, or morphology of the ECG at rest, such as complete left bundle branch block, 2nd and 3rd degree heart block, PR interval > 250 ms, etc.; c) Left ventricular ejection fraction (LVEF) < 50%; 8. Immunodeficiency diseases (HIV) and active hepatitis (hepatitis B virus [HBV], hepatitis C virus [HCV]), excluding carriers with asymptomatic chronic HBV or HCV. Active HBV, HCV, and HIV positive infection is defined as: d) HBsAg is positive and HBV DNA is ≥ 2000 cps/mL (or 500 IU/mL); e) HCV antibody is positive and HCV RNA is higher than the upper limit of normal (ULN) of the study site; f) HIV antibody is positive. 9. Diagnosed interstitial lung disease with or without symptoms, as well as conditions that may cause drug-induced lung toxicity or related pneumonia, or pulmonary symptoms that the investigator considers unsuitable for inclusion or high-risk factors that may lead to interstitial lung disease and are not suitable for inclusion.

  10. Subjects with other diseases that may affect the efficacy and safety of the study drug, including but not limited to:

  a) Active infection requiring antibiotic therapy within 14 days prior to the start of study treatment; b) Active autoimmune disease or a history of autoimmune disease, including but not limited to inflammatory bowel disease, autoimmune hepatitis, Guillain-Barré syndrome, demyelinating disease, extensive dermatitis, immune-related interstitial pneumonia, or Grave's disease requiring drug medication; c) History of primary immunodeficiency; d) Active pulmonary tuberculosis; 11. A large amount or symptomatic moderate amount of pleural effusion, pericardial effusion, ascites at screening, and the symptoms are poorly controlled after treatment such as paracentesis and drainage.

  12. Clinically significant gastrointestinal abnormalities or diseases at screening, resulting in great difficulties in drug intake, transport, or absorption (such as dysphagia, uncontrollable nausea and vomiting), etc.

  13. History of solid organ transplant. 14. Known or suspected allergy to the study drug or its analogues. 15. Pregnant and lactating women. 16. The investigators consider that the subjects are not suitable to participate in this study (e.g., the treatment is not in the best interest of the subjects, the subjects have poor compliance, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) events (for dose escalation phase) | up to 21 days following first dose
  DLT will be determined by definition during the DLT observation period.
Incidence and severity of adverse events(for dose escalation phase) | Until 30 days after the last dose or initiation of a new antineoplastic therapy, whichever occurs first
  The safety profile of HDM2006 will be assessed by monitoring the adverse events (AE) per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.
Change from baseline in HPK1 expression in tumor tissues (dose expansion) | through study completion, an average of 1 year
  HPK1 expression levels will be measured using Flow Cytometry. The unit of measure is percentage of positive cells.
Changes from baseline in pSLP-76 expression in tumor tissue (dose expansion) | From baseline through study completion, an average of 1 year
  pSLP-76 expression levels will be measured using Flow Cytometry. The unit of measure is percentage of positive cells.
Recommended Phase 2 Dose (RP2D) (for dose expansion phase) | through study completion, an average of 1 year
  The specific dose level of HDM2006 identified for use in the Phase 2 expansion phase

SECONDARY OUTCOMES:
Plasma concentration of HDM2006 | up to7 days following last dose
  Plasma concentration of HDM2006
Objective Response Rate (ORR)(for dose escalation phase) | through study completion, an average of 1 year
  Objective response rate (ORR), which includes best response of complete response (CR) or partial response (PR) as assessed by the investigator.
Time to Response (TTR) | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  TTR is defined as the interval from the start of study therapy to the first documentation of an objective response.
Progression free survival (PFS) | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  PFS is defined as the interval from the start of study therapy to the earlier of the first documentation of disease progression/relapse or death from any cause.
Duration of Response (DOR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to100 months
  DOR is defined as the interval from the first documentation of objective response to the earlier of the first documentation of disease progression/relapse or death from any cause.
Overall survival (OS) | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  OS is defined as the interval from the start of study therapy to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China